CLINICAL TRIAL: NCT02537587
Title: Effect of Varying the Protein and Dietary Fiber Content of Energy Bars on Their Glycemic and Insulinemic Impact
Acronym: Solstice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glycemic Index Laboratories, Inc (Industry)
Collaborators: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: GIL-1342; PEP-1324 (Other: PepsiCo)
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus
Keywords: Blood glucose; Blood insulin; Humans; Postprandial; Carbohydrate; Protein; Resistant starch; Sugar
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (7):
- Control 1 (Active Comparator): 67g of Control energy bar containing 4g protein, 15g fat, 42g carbohydrate, 2g fiber, and 24g sugar.
  Interventions: Other: Control 1
- Control 2 (Active Comparator): 86g of Control energy bar containing 5g protein, 20g fat, 55g carbohydrate, 3g fiber and 30g sugar
  Interventions: Other: Control 2
- 15/0 (Experimental): Experimental bar with 15% added resistant starch and 0% added protein; 66g portion containing 3g protein, 7g fat, 50g carbohydrate, 10g fiber and 16g sugar
  Interventions: Other: 15/0
- 15/0-LS (Experimental): Experimental bar with 15% added resistant starch and 0% added protein with reduced sugar; 84g portion containing 4g protein, 8g fat, 55g carbohydrate, 15g fiber and 15g sugar
  Interventions: Other: 15/0LS
- 15/5 (Experimental): Experimental bar with 15% added resistant starch and 5% added protein; 75g portion containing 9g protein, 7g fat, 52g carbohydrate, 12g fiber and 17g sugar
  Interventions: Other: 15/5
- 10/5 (Experimental): Experimental bar with 10% added resistant starch and 5% added protein; 72g portion containing 10g protein, 8g fat, 49g carbohydrate, 9g fiber and 19g sugar
  Interventions: Other: 10/5
- 10/10 (Experimental): Experimental bar with 10% added resistant starch and 10% added protein; 80g portion containing 17g protein, 7g fat, 49g carbohydrate, 9g fiber and 18g sugar
  Interventions: Other: 10/10

INTERVENTIONS:
Other: Control 1 — 67g of control bar
  Arms: Control 1
Other: Control 2 — 86g of control bar
  Arms: Control 2
Other: 15/0 — 66g of experimental bar 15/0
  Arms: 15/0
Other: 15/0LS — 84g of experimental bar 15/0LS
  Arms: 15/0-LS
Other: 15/5 — 75g of experimental bar 15/5
  Arms: 15/5
Other: 10/5 — 72g of experimental bar 10/5
  Arms: 10/5
Other: 10/10 — 80g of experimental bar 10/10
  Arms: 10/10

SUMMARY:
The purpose of this study was to determine the effect of changing the amounts of resistant starch, whey protein and sugar on the blood glucose and insulin responses elicited by energy bars. The investigators also compared the glucose and insulin responses to the rates at which the food bars were digested in-vitro (in the test tube). The investigators thought increasing resistant starch and reducing sugar would reduce the glucose and insulin responses, and that adding protein would reduce glucose and increase insulin. The investigators also thought the glucose and insulin responses in people would be related to the rate of digestion of the food bars in-vitro.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 20.0 to 34.9 kg/m²
* Fasting serum glucose <7.0mmol/L
* Non-smoker

Exclusion Criteria:

* Known to have diabetes
* Use of medications or presence of a medical condition considered by the principal investigator to increase risk to the participant or affect the results
* Known food allergy of any kind

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Incremental area under the blood glucose response curve | For 3 hours after consuming each test meal

SECONDARY OUTCOMES:
Incremental area under the serum insulin response curve | For 3 hours after consuming each test meal
Incremental area under the blood glucose response curve | For 2 hours after consuming each test meal
Incremental area under the serum insulin response curve | For 2 hours after consuming each test meal
Insulin:Glucose area under the curve ratio | For 3 hours after consuming each test meal
  Outcome 2 (incremental area under the insulin response curve for 3 hours) divided by Outcome 1 (incremental area under the glucose response curve for 3 hours)
Insulin:Glucose area under the curve ratio | For 2 hours after consuming each test meal
  Outcome 4 (incremental area under the insulin response curve for 2 hours) divided by Outcome 3 (incremental area under the glucose response curve for 2 hours)
Insulinogenic index | 30 minutes after consuming each test meal
  I30 divided by G30; where I30 is the serum insulin increment at 30 minutes and G30 is the blood glucose increment at 30 minutes; and where "increment" is defined as the concentration at 30 minutes minus the fasting concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — Glycemic Index Laboratories, Inc
Locations (1):
- Glycemic Index Laboratories, Inc., Toronto, Ontario, Canada

REFERENCES:
- [Derived] Wolever TM, van Klinken BJ, Bordenave N, Kaczmarczyk M, Jenkins AL, Chu Y, Harkness L. Reformulating cereal bars: high resistant starch reduces in vitro digestibility but not in vivo glucose or insulin response; whey protein reduces glucose but disproportionately increases insulin. Am J Clin Nutr. 2016 Oct;104(4):995-1003. doi: 10.3945/ajcn.116.132431. Epub 2016 Aug 31. PMID 27581470